CLINICAL TRIAL: NCT03817021
Title: ONE PATH: Optimizing Nutrition Education for Parents and Teachers for Healthy Growth
Acronym: ONE PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jennifer Savage Williams, Associate Professor of Nutritional Sciences, Penn State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DK120754-01 (NIH)
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-01

CONDITIONS: Childhood Obesity; Self-regulation; Appetite Regulation
Keywords: Responsive parenting; Early Childhood Education; Appetite Regulation
MeSH Terms: conditions — Pediatric Obesity; Self-Control | interventions — Appetite Regulation

STUDY DESIGN:
Intervention Model Description: Using Multiphase Optimization (MOST) Strategy, we will examine 3 treatment factors and their interactions to determine a 'best' or optimum approach to education of the Early Childhood Environment (ECE), child and family.
Masking Description: Parents, educators and children will not be informed of their treatment factor status, but it will not be hidden from them either.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- All Factors On (Experimental): ECE Provider intervention will be turned on Parent intervention will be turned on Child intervention will be turned on
  Interventions: Behavioral: ECE Provider; Behavioral: Parent Intervention; Behavioral: Child intervention
- ECE on/Parent on (Experimental): ECE Provider intervention will be turned on Parent intervention will be turned on Child intervention will be turned off
  Interventions: Behavioral: ECE Provider; Behavioral: Parent Intervention
- ECE on/Child on (Experimental): ECE Provider intervention will be turned on Parent intervention will be turned off Child intervention will be turned on
  Interventions: Behavioral: ECE Provider; Behavioral: Child intervention
- ECE on (Experimental): ECE Provider intervention will be turned on Parent intervention will be turned off Child intervention will be turned off
  Interventions: Behavioral: ECE Provider
- Parent on/Child on (Experimental): ECE Provider intervention turned off Parent intervention turned on Child intervention turned on
  Interventions: Behavioral: Parent Intervention; Behavioral: Child intervention
- Parent on (Experimental): ECE Provider intervention turned off Parent intervention turned on Child intervention turned off
  Interventions: Behavioral: Parent Intervention
- Child on (Experimental): ECE Provider intervention turned off Parent intervention turned off Child intervention turned on
  Interventions: Behavioral: Child intervention
- All Factors Off (No Intervention): ECE Provider intervention turned off Parent intervention turned off Child intervention turned off

INTERVENTIONS:
Behavioral: ECE Provider — Provide online training for Head Start educators
  Other Names: Responsive feeding for early childhood educators; ECE
  Arms: All Factors On; ECE on; ECE on/Child on; ECE on/Parent on
Behavioral: Parent Intervention — Coach parents remotely to educate them on responsive feeding and parenting
  Other Names: RF; Parent Responsive Feeding
  Arms: All Factors On; ECE on/Parent on; Parent on; Parent on/Child on
Behavioral: Child intervention — Through classrooms lessons cover 3 topics: 1) self-regulation, 2) hunger and fullness, and 3) mindfulness in eating and attention control practices
  Other Names: Appetite regulation; Child regulation
  Arms: All Factors On; Child on; ECE on/Child on; Parent on/Child on

SUMMARY:
This proposal uses an innovative methodological framework, the multiphase optimization strategy (MOST), to design an effective and efficient responsive feeding (RF) intervention that promotes child appetite self-regulation among a high-risk sample: families with preschoolers living in rural poverty. The principles of MOST emphasize efficiency, allowing identification of the most efficacious intervention components (i.e., components that contribute to treatment effects) while minimizing participant burden and cost. ONE PATH will intervene on ~768 dyads recruited from 56 classrooms serving largely low-income, rural populations.

DETAILED DESCRIPTION:
The ONE PATH: Optimizing Nutrition Education for Parents And Teachers for Healthy growth study will rigorously test the efficacy of responsive feeding (RF) and appetite regulation interventions. ONE PATH will intervene upon 3 unique targeted audiences, 1) Early Childhood Education providers (ECE), 2) preschool children, and 3) parents of the preschool children, to address childhood obesity in rural, under-served areas. ECE providers will receive online RF training and coaching. Preschool children will receive an experiential play-based curriculum delivered in the classroom focused on recognition of hunger and fullness cues and using attention control and mindfulness strategies to regulate food intake. Parents will receive RF and parenting guidance from ONE PATH educators through remote coaching. In addition to the three candidate interventions, all classrooms had the option to elect to participate in an existing evidence-based intervention (CORE intervention), the Nutrition and Physical Activity Self-Assessment of Child Care (Go NAP SACC) program. This component will not be tested as part of the optimized intervention.

Aim 1 is to identify which intervention components improve feeding practices and children's appetite regulation (primary), and BMI z-scores (secondary) over the 9-month school year. The 3 candidate intervention components include 1) RF interactive web-based training curriculum and coaching for ECE providers ("ECE provider intervention"), 2) classroom curriculum that teaches regulation strategies to preschool children ("child intervention"), and 3) responsive parenting (RP) curriculum and interactive activities for parents that provide opportunities to practice RF at home ("parent intervention"). The investigators will use the highly efficient multi-phase optimization (MOST) experimental strategy powered to detect main effects and all interactions.

Aim 2 is to improve understanding of the mechanisms by which the 3 candidate intervention components work, and determine if individuals respond differently to intervention components using the data from the experiment in Aim 1. The investigators will examine whether food security and child temperament explain the effects of the intervention on the outcomes (child appetite regulation, caregiver feeding practices, and child BMI z-score).

To investigate whether certain intervention components are more or less effective in certain subgroups, the investigators will explore moderation by child sex, race/ethnicity, and BMI categories.

ELIGIBILITY:
Inclusion Criteria:

* children must be enrolled in a participating Head Start or Pre-K Counts center
* children must be between 2 and 6 years old
* parent or primary caregiver must be 18 years or older
* parent/child English speaking
* ECE providers must be employed in participating Head Start or Pre-K Counts center

Exclusion Criteria:

* Parents will not be eligible to participate if their child is not eligible and/or not enrolled in the study
* ECE providers will not be eligible if they do not teach in a participating preschool classroom

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1461 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Child Appetite Regulation | Post intervention (~9 months)
  Difference in mean COMPX score at post-intervention between intervention and control conditions:
  Child appetite regulation skills will be assessed using the gold standard caloric compensation score (COMPX). On 2 occasions, children will be served a smoothie ~20 minutes prior to lunch - on 1 occasion, they will receive a low-calorie smoothie, and on the other a high-calorie smoothie (order will be randomized by classroom). Children will then be served an ad-libitum lunch (same foods on both occasions), and intake will be determined by pre- and post-weighing of food. The difference in intake between the two conditions reflects the child's ability to compensate for the higher calorie preload, a measure of appetite regulation. Caloric compensation score (COMPX) will be calculated as a percentage score. A COMPX of 100% reflects perfect caloric compensation. A COMPX higher than 100% indicates overcompensation, whereas a COMPX lower than 100% indicates under-compensation.
Parent feeding practices | Baseline and post intervention (~9 months)
  Differences in baseline-post change in parent feeding practice scores between intervention and control conditions
  Parent feeding practices will be assessed using the Structure and Control in Parent Feeding (SCPF) questionnaire, a 34-item measure that assesses positive, structure based feeding practices (i.e., limit-setting, consistent routines) and controlling feeding practices (i.e., restriction, pressure to eat). Items are scored on a 5-point likert scale (0 = never- 4 = always), with higher scores indicating higher frequency of engagement in a specific feeding behavior.
Parent feeding practices | Baseline and post intervention (~9 months)
  Differences in baseline-post change in parent feeding practice scores between intervention and control conditions. Parent feeding practices will be assessed using the Feeding to Manage Child Behavior questionnaire (FMCBQ), a 9-item measure that assesses parents' use of food to soothe and food as reward. Items are scored on a 5-point Likert scale (0 = never- 4 = always), with higher scores indicating higher frequency of engagement in food to soothe or as reward.
Early childhood educator (ECE) feeding practices | Post intervention (~9 months)
  Difference in percentage of educators engaging in specific feeding practices between intervention and control conditions at post-study.
  Early childhood educators feeding practices will be assessed using the Mealtime Observation in Childcare Checklist (MOCC). This measure will capture whether educators engage in specific feeding styles and practices during meal time. Some of the behaviors observed will include: whether educators pressured children to eat their food, praised children for trying a certain food or finishing their food, or if they provided food- or non-food related rewards to children for eating food. Additionally, we will observe how educators handled food refusal and if they supported children's self-regulation. For each item on the check list, observers indicate if they did or did not observe the behavior.
Parent feeding practices | Baseline and post intervention (~9 months)
  Differences in baseline-post change in parent feeding practice scores between intervention and control conditions
  Parent feeding practices will be assessed using the Caregiver's Feeding Styles Questionnaire (CFSQ), a 19-item measure which classifies caregivers into 1 of 4 feeding styles (authoritarian, authoritative, indulgent and uninvolved). Items are scored on a 5-point scale (1=never-5=always), with higher scores indicating higher frequency of engagement in a specific feeding style.

SECONDARY OUTCOMES:
BMI z-scores | Baseline and post intervention (~9 months)
  Difference in change in BMI z-scores from baseline to post between intervention and control conditions
  Children's weights and heights will be obtained at baseline and the end of the study using standard procedures. BMI will be calculated and values will be standardized to z-scores and percentiles according to Centers for Disease Control (CDC) standards and adjusted for child's sex and age.
Child Appetite Regulation and Satiety Responsiveness | Baseline and post intervention (~9 months)
  Differences in change from baseline-post intervention in calories consumed in the Eating in the Absence of Hunger (EAH) task between intervention and control conditions.
  The EAH procedure measures children's snack food consumption when not hungry. Children will be presented with a variety of snack foods shortly after being fed a full meal. The snacks will be weighed prior to and following the procedure to calculate intake. This will be evaluated at baseline and post intervention.
Child Appetite Regulation and Satiety Responsiveness | Baseline and post intervention (~9 months)
  Differences in change in appetitive traits (parent-rated) from baseline-post, and mean appetitive traits at post-intervention (ECE provider-rated) between intervention and control conditions.
  Child appetitive traits will be assessed using the Children's Eating Behavior Questionnaire, which will be completed by parents at baseline and post intervention and by ECE providers post intervention only. This measure assesses children's eating style using a 5-point scale (1 = never - 5 = always).
Classroom/school food environment | Post intervention (~9 months)
  Differences in percent of classrooms exhibiting specified characteristics of food environment at post-intervention between intervention and control conditions.
  The ECE environment, including food and beverages served, physical environment, teacher engagement, and feeding practices will be assessed observationally at baseline (subset) and the conclusion of the project (all classrooms) using the validated MOCC. We hope to observe more teacher engagement, positive environment, and feeding practices in the classrooms post-intervention.
Waist Circumference | Baseline and post intervention (~9 months)
  Differences in mean waist circumference at post-intervention between intervention and control conditions. Waist circumference values will be standardized to z-scores and percentiles according to sex- and age-specific guidelines. Waist circumference will be obtained using standardized procedures at baseline and post-intervention.
Weight Status | Post intervention (~9 months)
  Differences in percentage of overweight and obesity status (compared to not having overweight or obesity) at post-intervention between intervention and control conditions.
  BMI percentiles according to Centers for Disease Control (CDC) standards and adjusted for child's sex and age will be calculated and use to determine prevalence of overweight (≥ 85th percentile) and obesity (< 95th percentile).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Williams, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be available to researchers on request after the conclusion of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available one year following the conclusion of the study.
Access Criteria: Researchers must submit a request with planned use to the PI, and complete a data sharing agreement with Penn State University.